CLINICAL TRIAL: NCT03484247
Title: Injection Optimization of Infraclavicular and Axillary Brachial Plexus Block: Comparison of Number of Attempts and Performance Time
Brief Title: Injection Optimization of Infraclavicular and Axillary Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Sevtap Cemaloglu, Principal Investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: sevtap 1
Record Dates: First submitted 2018-03-12; First posted 2018-03-30 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Brachial Plexus Block
Keywords: infraclavicular block; axillary block

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Infraclavicular (Active Comparator): Infraclavicular Brachial Plexus Block: The inferolateral of the subclavian artery will be targeted with a 85 mm peripheral nerve stimulator needle with ultrasound guidance. When the needle tip was seen near the posterior cord of brachial plexus local anesthetic will be administered with single injection after aspiration.
  Interventions: Other: Infraclavicular brachial plexus block
- Group Axillary (Active Comparator): Axillary Brachial Plexus Block: The procedure will be performed with a 50 mm peripheral nerve stimulator needle with ultrasound guidance. Local anesthetic will be administered with multiple injection (radial, ulnar, median and musculocutaneous nerves) after aspiration.
  Interventions: Other: axillary brachial plexus block

INTERVENTIONS:
Other: Infraclavicular brachial plexus block — Infraclavicular block will be performed with ultrasound guidance and peripheric nerve stimulator. Local anesthetic will be administered after aspiration, via peripheric nerve needle according to mentioned technique ( https://www.nysora.com/)
  Arms: Group Infraclavicular
Other: axillary brachial plexus block — Axillary nerve block will be performed with ultrasound guidance and peripheric nerve stimulator. Local anesthetic will be administered after aspiration via peripheric nerve needle according to mentioned technique ( https://www.nysora.com/)
  Arms: Group Axillary

SUMMARY:
In upper extremity surgery, brachial plexus block (BPB) is routinely applied successfully as general anesthesia (GA). However, BPB is less invasive technique than GA. Peripheral nerve blocks have some potential benefits, such as lower risk of nausea and vomiting, early ambulation, early discharge, and better control of postoperative pain. The BPB is applied to various areas such as axillary, supraclavicular, infraclavicular and interscalene areas under the guidance of ultrasound and nerve stimulator. Among these methods, BPB administration success rates are around 95-100%. The other condition is anesthetic time which is important for the turnover of operating room. Anesthetic time is the sum of the performance time and onset time. In addition performance time and number of needle attempts also associated with patient satisfaction. The primary aim of this study is to determine the number of attempts and the performance time with the onset time and anesthetic time. If the procedure is simple, the performance time may be shorter. Therefore, the investigators aim that comparison of two different procedures which are single injection infraclavicular brachial plexus block and multiple injection axillary brachial plexus block by ultrasound guidance. In addition, the investigators will examine the duration of anesthesia and surgery, the duration of sensory and motor block endings, patient comfort and pain scales in the postoperative period.

DETAILED DESCRIPTION:
60 participants who underwent forearm or hand surgery with the axillary or infraclavicular brachial plexus block method and who have an American Society of Anesthesiologists physical status classification (ASA) score of I-II-III between the ages of 18-75 will be followed up. Number of needle attempts, block performance time, sensorial and motor block onset time, total anesthetic time, surgical duration, duration of sensory block formation, and duration of motor block formation will be evaluated with the information obtained from participants with axillary block or infraclavicular block. After surgery, participants satisfaction, visual analogue scales (VAS), sensory block ending times, motor block ending times and first analgesic requirement time will be assessed at postoperative 2. -8. -12. -24. hours by physical examination and questions. As a result of these evaluations, both groups will be compared statistically. (After the patients are informed in detail, the volunteer certificate will be obtained from the patients who agree to participate in the study.)

ELIGIBILITY:
Inclusion Criteria:

* Axillary or infraclavicular brachial plexus block who underwent forearm or hand surgery
* ASA score I-II-III
* Body weight> 45 kg or BMI <40 kg / m2

Exclusion Criteria:

* Under 18 years old or over 75 years old
* Body weight <45 kg or BMI> 40 kg / m2
* ASA score above III
* Pregnant or lactating
* Coagulopathy or anticoagulant medication
* Allergies about using local anesthetic drugs
* Neurological deficit
* Renal insufficiency or liver failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
time to brachial plexus block performance | from the first second of brachial plexus imaging with ultrasound until the needle remove from the skin will be assessed up to ten minutes
  performance time will hold with a stopwatch

SECONDARY OUTCOMES:
number of needle attempt | during the procedure
  number of needle attempt will be count during the procedure
time to brachial plexus block onset | after end of the procedure 5th, 10th, 15th, 20th, 25th, 30th minutes
  nerves will have sensorial and motor examination

OTHER OUTCOMES:
patient satisfaction | 5 minutes after the operation
  patients will answer the question that 'how would you rate your satisfaction of procedure?'
  0:poor, 1:good, 2:excellent

CONTACTS AND LOCATIONS:
Locations (1):
- Diskapi TRH, Ankara, Turkey (Türkiye)